CLINICAL TRIAL: NCT05209425
Title: Pharmacokinetics Evaluation of Different Vitamin D3 Formulations
Brief Title: Pharmacokinetics Evaluation of Vitamin D Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Factors Group of Nutritional Companies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-11-001
Record Dates: First submitted 2021-12-20; First posted 2022-01-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Vitamin D
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: parallel, randomized blinded study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Regular Vitamin D3 1000IU (Active Comparator): The first group receives regular Vitamin D3 1000IU
  Interventions: Dietary Supplement: Vitamin D3
- Microencapsulated Vitamin D3 1000IU (Active Comparator): The second group receives microencapsulated Vitamin D3 1000IU
  Interventions: Dietary Supplement: Vitamin D3
- Regular Vitamin D3 2500IU (Active Comparator): The third group receives regular Vitamin D3 2500IU
  Interventions: Dietary Supplement: Vitamin D3
- Microencapsulated Vitamin D3 2500IU (Active Comparator): The fourth group receives microencapsulated Vitamin D3 2500IU
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Participants are randomly divided into 4 groups. The first group receives regular Vitamin D3 (1000IU), the second receives microencapsulated D3 (1000IU), the third group receives regular Vitamin D3 (2500IU), the fourth receives microencapsulated D3 (2500 IU). Plasma concentrations of Vitamin D (D3, 25(OH)D3 and D2) are measured at baseline-before treatment start (day 0), during treatment (day 14) and at end of treatment (day 30). After the end of supplementation, blood vitamin D concentrations are checked again at day 45 and day 60.

SUMMARY:
The primary objective of this study is to evaluate plasma concentrations of Vitamin D (25-hydroxyvitamin D; 1,25-dihydroxyvitamin D) of different Vitamin D formulations in healthy volunteers at two concentrations. Pharmacokinetic parameters (Serum 25(OH)D and 1,25(OH)2D ng/ml) are compared with those of a regular Vitamin D formulation and a new (microencapsulated) LipoMicel Vitamin D formulation.

The secondary objective of this study is to evaluate safety blood parameters- The following blood parameters (serum levels) are checked: Alkaline Phosphatase, ALT, AST, Bilirubin, CRP, Creatinine, GGT. In addition, mineral levels-such as calcium, magnesium and phosphorus, potassium and sodium-are measured before and at the end of the study.

DETAILED DESCRIPTION:
Study Design:

At least 40 healthy volunteers of both sexes in the age range 21-65 participate in a parallel, randomized blinded study conducted with different vitamin D3 products.

Each treatment is administered orally per day at a total dose of 1000 UI and 2500 IU vitamin d3 (cholecalciferol), together with breakfast, over a period of 30 days.

Participants are randomly divided into 4 groups (at least 10 per group):

The first group receives regular Vitamin D (1000IU), the second receives microencapsulated D3 (1000IU), the third group receives regular Vitamin D (2500IU), the fourth receives microencapsulated D3 (2500 IU).

Plasma concentrations (serum levels) of Vitamin D (25(OH)D and 1,25(OH)2D ng/ml are measured at baseline-before treatment start (day 0), during treatment (day 5, 10 and 15; one blood collection per day) and at end of treatment (day 30).

After the end of supplementation, blood vitamin D concentrations are checked again at day 45 and day 60.

The entire study session will span the course of 60 days. Participants are asked to attend 7 visits at LifeLabs to collect venous blood samples.

Each Vitamin D treatment is consumed with a glass of water along with breakfast for a period of 30 days.

Safety blood work is performed upon study enrolment, at the end of the Vitamin supplementation (day 30)- and at the end of the study (day 60) at Life Labs.

The following blood parameters are checked and must be within normal ranges to participate the study: Alkaline Phosphatase, ALT, AST, Bilirubin, CRP, Creatinine, GGT.

Mineral levels-such as calcium, magnesium and phosphorus-are measured before and at the end of the study (day 30).

All participants must understand written and spoken English and give written informed consent before any study speciﬁc procedure will be carried out.

All tested products are formulation manufactured by Factors Group.

ELIGIBILITY:
Inclusion Criteria:

* age between 21 and 65 years; avoid consumption of any additional food supplements containing vitamin D; avoid use of tanning beds or other artificial UVB sources.

Participants must complete an online questionnaire on their medical history, weight, height, lifestyle (smoking, exercising etc.) and dietary habits relating to food rich in vitamin D, including other dietary supplementations.

Exclusion Criteria:

* use of vitamin D, calcium, magnesium, fish oil, or omega 3 fatty acids supplements; history of acute or chronic illness (such as gastrointestinal, liver and kidney disorders, osteoporosis …); pregnancy or lactation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Vitamin D serum level: change of 1,25-Dihydroxyvitamin D | at day 0 (before treatment), at day 5, 10, 15 (during treatment), at day 30 (end of treatment), at day 45 and 60 (after treatment).
  Venous blood samples are collected to measure concentrations of 1,25-Dihydroxyvitamin D
Evaluation of Vitamin D serum level: change of 25-Hydroxyvitamin D | at day 0 (before treatment), at day 5, 10, 15 (during treatment), at day 30 (end of treatment), at day 45 and 60 (after treatment).
  Venous blood samples are collected to measure concentrations of 25-Hydroxyvitamin D

SECONDARY OUTCOMES:
Safety blood work evaluation - change of aspartate aminotransferase (AST) | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of AST
Safety blood work evaluation - change of alanine aminotransferase (ALT) | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of ALT
Safety blood work evaluation - change of alkaline phosphatase | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of alkaline phosphatase
Safety blood work evaluation - change of bilirubin | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of total bilirubin
Safety blood work evaluation - change of gamma-glutamyl transferase (GGT) | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of GGT
Safety blood work evaluation - change of creatinine | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of creatinine
Safety blood work evaluation - change of C Reactive Protein (CRP) | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of CRP
Safety blood work evaluation - change of mineral levels such as calcium | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of calcium
Safety blood work evaluation - change of mineral levels such as magnesium | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of magnesium
Safety blood work evaluation - change of mineral levels such as phosphate | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of phosphate
Safety blood work evaluation - change of mineral levels such as sodium | at day 0 (before treatment), at day 30 (end of treatment), at day 60 (after treatment).
  Venous blood samples are collected to measure concentrations of sodium

CONTACTS AND LOCATIONS:
Locations (1):
- Natural Factors, Coquitlam, British Columbia, Canada

REFERENCES:
- [Derived] Solnier J, Chang C, Zhang Y, Kuo YC, Du M, Roh YS, See J, Brix J, Gahler RJ, Green T, Wood S. A Comparison and Safety Evaluation of Micellar versus Standard Vitamin D3 Oral Supplementation in a Randomized, Double-Blind Human Pilot Study. Nutrients. 2024 May 22;16(11):1573. doi: 10.3390/nu16111573. PMID 38892507